CLINICAL TRIAL: NCT03242382
Title: Phase II Multicenter Trial of Palbociclib in Second Line of Advanced Sarcomas With CDK4 Overexpression.
Brief Title: Trial of Palbociclib in Second Line of Advanced Sarcomas With CDK4 Overexpression.
Acronym: PalboSarc
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS-51
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Soft-tissue Sarcoma; Osteosarcoma; Chordoma
Keywords: advanced; sarcoma; cdk4
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Chordoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbocilib (Experimental): Palbociclib will be administered orally at a dose of 125 mg once a day for 21 consecutive days followed by 7 rest days to comprise a complete cycle of 28 days.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision
  Other Names: Ibrance

SUMMARY:
Non-randomized, open, two-cohort, phase II, multicenter national clinical trial. 20 sites in Spain.

Cohort 1 includes soft-tissue sarcoma and osteosarcoma (21 patients), while Cohort 2 includes chordoma patients only (19 patients).

Palbociclib will be administered orally at a dose of 125 mg once a day for 21 consecutive days followed by 7 rest days to comprise a complete cycle of 28 days. Treatment will continue until disease progression, development of unacceptable toxicity, non-compliance, withdrawal of consent by the patient or investigator decision.

The main goal is to determine progression-free survival rate (PFSR) according to RECIST 1.1 at 6 months.

ELIGIBILITY:
Inclusion Criteria (Cohort 1: STS and osteosarcoma):

1. Over-expression of CDK4 (mRNA expression) and a low-to-normal p16 expression (mRNA expression) measured in paraffin embedded tumor samples at study entry.
2. ECOG 0-1 at enrollment.
3. Diagnosis of soft tissue sarcoma or osteosarcoma (in both cases with metastasis or locally advanced, unresectable).
4. Disease progression documented within 6 months prior to study entry.
5. Patients must have the following laboratory results:

   * ANC ≥ 1,500/mm3 (1.5 x 109/L);
   * Platelets ≥ 100,000/mm3 (100 x 109/L);
   * Hemoglobin ≥ 9 g/dL (90 g/L);
   * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 60 mL/min;
   * Total serum bilirubin ≤ 1.5 x ULN (≤ 3.0 x ULN if Gilbert's disease);
   * AST and/or ALT ≤ 3 x ULN (≤ 5.0 x ULN if liver metastases present);
   * Alkaline phosphatase ≤ 2.5 x ULN (≤ 5.0 x ULN if bone or hepatic metastasis present);
6. Patients must have signed written informed consent to participate in the clinical study, and to provide at least two paraffin embedded tumor blocks for the molecular analyses at screening stage.
7. Biopsy at baseline if there are no archived tumor samples obtained within 3 months prior to treatment initiation.
8. Patients must have received standard treatments for at least one, two or three lines for advanced disease.
9. Age between 18 and 80 years (both ages included).
10. Measurable disease according to RECIST 1.1 criteria.
11. All patients (men and women) in fertile age must use an effective contraception method during the entire treatment with palbociclib and for at least 90 days after the last dose. Pregnancy must be ruled out through urine or blood test (negative pregnancy test) for the inclusion in the study. Men must be informed to consider spermatic preservation before treatment initiation due to infertility risks.

Exclusion Criteria (Cohort 1: STS and osteosarcoma):

1. Previous treatment with any anti CDK4 or immune checkpoint inhibitor.
2. Diagnosis of Ewing sarcoma or rhabdomyosarcoma.
3. Diagnosis of well differentiated/dedifferentiated liposarcoma.
4. Patients irradiated on the only target lesion available.
5. Patients having received more than three lines for advanced disease.
6. History of other neoplastic disease with the exception of basal cell carcinoma or in situ cervical cancer adequately treated.
7. Serious cardiovascular disease (NYHA >= 2)
8. Grade 3 or superior toxicity according to CTCAE 4.0 if the investigator considers this can significantly interfere in the toxicity of the drug under study.
9. Patients not recovered from a previous toxicity to at least CTCAE Grade 1 due to prior chemotherapy, radioactive, or biological cancer therapy (including monoclonal antibodies).
10. Patients not recovered from minor or major surgery or having undergone a major surgery within the last 4 weeks prior to initiation of study treatment.
11. Central nervous system metastasis.
12. Pregnant or breastfeeding patients, or those expecting to conceive or father children within the projected duration of treatment.
13. Foods or drugs known as CYP3A4 inhibitors/inducers; CYP3A4 substrates with narrow therapeutic windows, or known to prolong QTc interval.
14. Major surgery, chemotherapy, radiotherapy, any agent under investigation, or other antineoplastic therapy within 4 weeks prior to inclusion. Patients having received a previous radiotherapy ≥25% of bone marrow are not eligible, regardless of when it was received.
15. QTc > 480 ms; personal or family history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsades de Pointes (TdP).
16. Any of the following situations within 6 months prior to study drug administration: myocardial infarction, serious/unstable angina, current cardiac dysrhythmias Grade ≥ 2 NCI-CTCAE version 4.0, atrial fibrillation of any grade, bypass graft in coronary/peripheral artery, symptomatic congestive cardiac failure, cerebrovascular accident including transient ischemic attack, or symptomatic pulmonary embolism.
17. Known hypersensitivity to any PD 0332991 or excipients.
18. Active or recent suicide attempt or behavior.

Inclusion Criteria (Cohort 2: Chordomas):

1. Mutation of CDKN2A gen.
2. ECOG 0-1 at the time of inclusion.
3. Centrally confirmed diagnosis of chordoma (metastatic or locally advanced inoperable).
4. Disease progression according to RECIST 1.1, within the year prior to inclusion, to previous treatment (surgery, radiotherapy or systemic treatment).
5. Patients are not candidates for salvage surgery or radiotherapy at the time of inclusion.
6. Patients must have the following lab results:

   * Absolute neutrophil count ≥ 1,500/mm3 (1.5 x 109/L);
   * Platelets ≥ 100,000/mm3 (100 x 109/L);
   * Hemoglobin ≥ 9 g/dL (90 g/L);
   * Blood creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 60 mL/min;
   * Total blood bilirubin ≤ 1.5 x ULN (≤ 3.0 x ULN if Gilbert's disease);
   * AST and/or ALT ≤ 3 x ULN (≤ 5.0 x ULN if there is liver metastasis);
   * Alkaline phosphatase ≤ 2.5 x ULN (≤ 5.0 x ULN if there is bone or liver metastasis);
7. The patients must have signed the written consent to participate in the clinical study, and to provide the tumor blocks in paraffin for the molecular analysis of the screening phase.
8. Biopsy at baseline if there are no archive tumor samples obtained in the 3 months prior to starting treatment. If there are tumor samples within this period, there should not be subsequent treatments.
9. Patients may have received up to 3 previous lines of systemic treatment.
10. Age between 18 and 80 years (both ages included).
11. Measurable disease according to RECIST 1.1 criteria.
12. All patients (male and female) of childbearing potential must use effective contraception throughout treatment with palbociclib and for at least 90 days after the last dose. Pregnancy must be ruled out by urine or blood test (negative pregnancy test) for inclusion in the study. Men should be told to consider sperm preservation before starting treatment due to the risks of infertility.

Exclusion Criteria (Cohort 2: Chordomas):

1. Prior treatment with any anti-CDK4 or immune checkpoint inhibitors.
2. Diagnosis other than chordoma according to central review.
3. Patients irradiated in the only available target lesion.
4. Patients who have received more than three lines for advanced disease.
5. History of other neoplastic disease with the exception of adequately treated basal cell carcinoma or cervical cancer in situ. This criterion will be individually assessed with the research team.
6. Severe cardiovascular disease (NYHA >= 2).
7. Grade 3 toxicity or higher according to CTCAE 5.0 if, in the investigator's opinion, it can significantly interfere with the toxicity of the drug under study.
8. Patients who have not recovered from previous toxicity up to CTCAE grade 1 due to previous antineoplastic treatment with chemotherapy, radiotherapy, or biological therapy (including monoclonal antibodies).
9. Patients who have not recovered from minor or major surgery or who have had major surgery within 4 weeks prior to the start of study treatment.
10. Metastases in the central nervous system.
11. Patients who are pregnant or lactating, or who expect to conceive children during the treatment period.
12. Foods or drugs known to be inhibitors/inducers of CYP3A4; CYP3A4 substrates with narrow therapeutic windows, or known to prolong the QTc interval.
13. Major surgery, chemotherapy, radiation therapy, any investigational agent, or other antineoplastic therapy within 4 weeks prior to enrollment. Patients who have received prior radiation therapy to ≥25% of the bone marrow are not eligible, regardless of when received.
14. QTc > 480 ms; personal or family history of long or short QT syndrome, Brugada syndrome, or known history of QTc prolongation, or Torsades de Pointes (TdP).
15. Any of the following within 6 months prior to study drug administration: Myocardial infarction, severe/unstable angina, current NCI-CTCAE version 5.0 Grade ≥ 2 cardiac dysrhythmias, any grade atrial fibrillation, implant coronary/peripheral artery pacemaker, symptomatic congestive heart failure, cerebrovascular accident including transient ischemic attack, symptomatic pulmonary embolism, or interstitial lung disease (ILD).
16. Known hypersensitivity to any PD 0332991 or excipients.
17. Active or recent suicidal intent or behavior.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate | At 6 months
  Efficacy measured through the progression free survival (PFS) rate at 6 months, evaluated with RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 months
  Efficacy measured through the overall response rate (ORR) (complete response [CR] and partial response [PR]), evaluated with RECIST 1.1 criteria. The evaluation criteria will be based on the identification of target lesions in baseline and their follow-up until tumor progression.
Efficacy measured through response according to Choi criteria measured through response according to Choi criteria: | 6 months
  Efficacy measured through response according to Choi criteria. The evaluation criteria will be based on the identification of target lesions in baseline and their follow-up until tumor progression.
Efficacy measured through median PFS | 6 months
  Efficacy measured through median PFS.
Efficacy measured through PFS rate at 3 months | 3 months
  Efficacy measured through PFS rate at 3 months.
Overall survival (OS) | 2 years
  Overall survival (OS) measured from the date of treatment initiation with palbociclib until date of death, whichever the cause.
Clinical Benefit Rate (CBR) | 6 months
  Clinical Benefit Rate (CBR). Patients having shown complete response, partial response, or disease stabilization during 6 months or more, showing clinical improvement symptoms, will be considered as having experienced clinical benefit.
Palbociclib safety profile | 1 year
  Palbociclib safety profile, through the evaluation of adverse events (type, incidence, severity, timing of appearance, related causes) observed in physical explorations and laboratory tests. Toxicity will be assessed and tabulated using NCI-CTCAE 4.0 (first cohort; STS and osteosarcoma) and 5.0 (second cohort; chordomas).

CONTACTS AND LOCATIONS:
Overall Officials: Irene Carrasco García, MD, Study Director — Hospitales Universitarios Virgen del Rocío; Roberto Díaz, MD, Study Director — Hospital Universitario La Fe; Javier Martínez Trufero, MD, Principal Investigator — Hospital Miguel Servet; Yolanda Vidal, MD, Principal Investigator — Complejo Hospitalario Universitario de Santiago; Juan Luís García Llano, MD, Principal Investigator — Hospital Universitario Central de Asturias; Antonio López-Pousa, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Diego Jara, MD, Principal Investigator — Hospital Universitario 12 de Octubre; Isabel Sevilla, MD, Principal Investigator — Hospital Universitario Virgen de la Victoria; Javier Martín Broto, Principal Investigator — Hospital Universitario Fundación Jiménez Díaz; Anna Estival, Principal Investigator — Germans Trias i Pujol Hospital; Luís Miguel de Sande, Principal Investigator — Complejo Asistencial Universitario de León; Rosa Álvarez, Principal Investigator — Hospital General Universitario Gregorio Marañón; Claudia Valverde, Principal Investigator — Hospital Universitari Vall d'Hebrón; Andrés Redondo, Principal Investigator — Hospital Universitario La Paz; Josefina Cruz, Principal Investigator — Hospital Universitario de Canarias; Javier Lavernia, Principal Investigator — Instituto Valenciano de Oncología; Pablo Luna, Principal Investigator — Hospital Son Espases; Jerónimo Martínez, Principal Investigator — Hospital Universitario Virgen de la Arrixaca; Xavier García del Muro, Principal Investigator — Institut Català d'Oncología l'Hospitalet; Antonio Casado, Principal Investigator — Hospital San Carlos, Madrid
Locations (19):
- Spain (19):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Institut Català d'Oncología l'Hospitalet, Barcelona
  - Complejo Asistencial Universitario de León, León
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided